CLINICAL TRIAL: NCT05179434
Title: A Randomized Clinical Study of Retrograde Reperfusion of Renal Graft to Reduce Ischemic-Reperfusion Injury
Brief Title: A Study of Retrograde Reperfusion of Renal Graft to Reduce Ischemic-reperfusion Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West Kazakhstan Medical University (Other)
Responsible Party: Principal Investigator, Myltykbay Rysmakhanov, PhD-doctoral, Department of Surgery No 2, MD, West Kazakhstan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 116.23.11.2020
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Kidney Transplantation; Ischemic Reperfusion Injury; Reperfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde graft reperfusion (Experimental): Kidney transplantation with retrograde venous reperfusion of renal graft followed by arterial reperfusion
  Interventions: Procedure: Retrograde renal graft reperfusion
- conventional antegrade perfusion (Active Comparator): Kidney transplantation with conventional arterial reperfusion of renal graft (without retrograde venous reperfusion)
  Interventions: Procedure: Conventional antegrade renal graft reperfusion (without retrograde reperfusion)

INTERVENTIONS:
Procedure: Retrograde renal graft reperfusion — Retrograde venous reperfusion of the renal graft during the kidney transplant procedure with consequent arterial reperfusion
  Other Names: Venous reperfusion
  Arms: Retrograde graft reperfusion
Procedure: Conventional antegrade renal graft reperfusion (without retrograde reperfusion) — Conventional arterial antegrade renal graft reperfusion during the kidney transplant procedure
  Other Names: Arterial reperfusion
  Arms: conventional antegrade perfusion

SUMMARY:
To evaluate whether retrograde venous reperfusion of a renal graft before antegrade arterial reperfusion can reduce ischemic-reperfusion injury.

All registered eligible candidates for kidney transplant will be randomized to receive either:

* retrograde venous, then arterial reperfusion or
* antegrade arterial reperfusion.

DETAILED DESCRIPTION:
According to our hypothesis, retrograde venous reperfusion prevents and reduces the immediate and long-term effects of renal allograft ischemic-reperfusion injury.

For the study Chi-square method of sample size estimation with a=0,05, b=0,20 required a 14 subject per group.

The study will include 30 potential kidney recipients for both group aged 18-60 years who will receive kidney transplants. Only adult patients undergoing primary living donor kidney transplantation with standard three-component immunosuppression will be enrolled to the study.The main study group will consist of 15 patients with retrograde graft reperfusion, and control group - will include 15 kidney recipients with only conventional antegrade arterial reperfusion (without retrograde reperfusion).

Patients of the study group with standard kidney implantation surgery will undergo retrograde reperfusion through the renal vein after venous anastomosis. After the venous anastomosis of the graft, an arterial anastomosis is applied with the renal artery without tightening the suture to leave a lumen sufficient for the outflow of retrograde blood. Then the retrograde blood flow through the renal vein is started, venous blood fills the graft and flows through the renal artery through the lumen of the anastomosis in a volume of 80-100 ml. Retrograde blood collected for gas and lactate analysis at the beginning of reperfusion, at the first minute and at the fifth minute. Further, the sutures of the arterial anastomosis are tightened, and after tying, a typical antegrade reperfusion of the graft through the renal artery is performed.

Patients in the control group will undergo standard kidney implantation surgery with typical antegrade arterial reperfusion.

T-test and Mann-Whitney test will be used to compare the median of urea, creatinine levels in serum and glomerular filtration rate (GFR) on the 1st, 7th, 14th, 30th, 60th postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage kidney disease who are ready for kidney transplantation;
* Panel reactive antibodies (PRA) less than 20%.
* informed consent to participate in the study.

Exclusion Criteria:

* recipients preparing for combined organ transplantation;
* recipients with previously performed transplantation of another organ;
* recipients preparing for transplantation with a different immunosuppressive regimen;
* upcoming blood group incompatibility (AB0-i) transplant;
* PRA antibodies more than 20%;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Renal graft and recipients survival | 3 months
  Renal graft function quality and recipients survival

SECONDARY OUTCOMES:
Median serum creatinine levels | 1 months
  Normalization of creatinine levels in dynamics
Median serum urea levels | 1 months
  Normalization of serum urea levels in dynamics
Median glomerular filtration rate (GFR) levels | 1 month
  Normalization of glomerular filtration ratio (GFR) in dynamics

CONTACTS AND LOCATIONS:
Locations (1):
- West Kazakhstan Medical University, Aktobe, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tasoulis MK, Douzinas EE. Hypoxemic reperfusion of ischemic states: an alternative approach for the attenuation of oxidative stress mediated reperfusion injury. J Biomed Sci. 2016 Jan 19;23:7. doi: 10.1186/s12929-016-0220-0. PMID 26786360
- [Background] Molacek J, Opatrny V, Matejka R, Baxa J, Treska V. Retrograde Oxygen Persufflation of Kidney - Experiment on an Animal. In Vivo. 2016 11-12;30(6):801-805. doi: 10.21873/invivo.10997. PMID 27815464